CLINICAL TRIAL: NCT02242539
Title: Tools to Improve Parental Recognition of Developmental Deficits in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: Harvard University (Other); Innovations for Poverty Action (Other)
Responsible Party: Principal Investigator, Peter Rockers, Assistant Professor, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14-2948
Record Dates: First submitted 2014-09-12; First posted 2014-09-17 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Malnutrition; Child Development
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Height measurement poster (Experimental)
  Interventions: Behavioral: Height measurement poster
- Community-based monitoring (Experimental)
  Interventions: Behavioral: Community-based monitoring
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Height measurement poster — Each household is provided with a poster which study personnel help to hang on the wall. The poster clearly indicates height-for-age benchmarks and stunting cut-offs for study-age children. Parents are provided training on how to measure their children at regular intervals, and interpret height readings to determine whether their child is developing normally or is stunted.
  Arms: Height measurement poster
Behavioral: Community-based monitoring — Once every three months, villages are visited by study staff who measure children's heights and weights, and parents are informed if their children are below the reference measures established by the World Health Organization. If a child's weight is such that the child is classified as severely malnourished, the child is referred to the nearest health center for treatment. If the child is stunted (height-for-age z-score more than 2 standard deviations below the reference median), we provide parents with a supply of "Yummy Soy" powder, a fortified soy and maize mix popular among parents and widely available in local super markets. Parents are instructed to give one or two tea spoons of the mix to the child each day.
  Arms: Community-based monitoring

SUMMARY:
In this study, we aim to improve child nutrition by increasing parents' awareness of their children's physical growth. We use a cluster-randomized trial design to evaluate two interventions that provide parents with regular information on their children's physical development and growth: 1) distribution of full-sized growth charts for measurement of child height within households; and 2) organization of community-based meetings, during which children's height and weight are measured by trained project staff.

DETAILED DESCRIPTION:
The target population for the study will be children between the ages of 6 and 18 months at baseline living in small-scale farming households in Chipata District, Zambia. As part of a cluster-randomized trial titled "Food Constraints, Yield Uncertainty and 'Ganyu' Labor" funded by IZA-DFID (PI: G Fink), 3,100 farming households in approximately 180 rural villages in Eastern Province are currently enrolled in a two-year study, which aims at assessing the effect of food loan programs on agricultural productivity. The study described here uses the "Food Constraints" population as a sampling frame; all households enrolled in the "Food Constraints" program that have a child between 6 and 18 months are invited to participate in this add-on trial. We anticipate that there will be around 600 eligible households recruited for this study. Study duration is about 18 months. Selected households will be visited for study enrollment and a short baseline assessment in September 2014, at which time the two interventions will also be rolled out. Final impact of the interventions will be assessed one year later, in September 2015.

ELIGIBILITY:
Inclusion Criteria:

* All households with a child between the ages of 6 and 18 months at baseline

Exclusion Criteria:

* None

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 547 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Height-for-age z-score | At the end of one year
  Children's heights will be measured and height-fore-age z-scores will be determined using standards published by the World Health Organization
Child development outcomes | At the end of one year
  Through parental reports and child tasks we will measure various aspects of child development, including motor skills and verbal skills

SECONDARY OUTCOMES:
Mid-upper arm circumference (MUAC) | At the end of one year
  Children will be measured for mid-upper arm circumference (MUAC) using standard measurement strips
Dietary intake | At the end of one year
  Parents will be asked to report on children's dietary intake during the day preceding the survey

CONTACTS AND LOCATIONS:
Overall Officials: Günther Fink, PhD, Principal Investigator — Harvard University; Peter Rockers, ScD, Principal Investigator — Boston University
Locations (1):
- Household sample, Chipata District, Zambia

REFERENCES:
- [Derived] Fink G, Levenson R, Tembo S, Rockers PC. Home- and community-based growth monitoring to reduce early life growth faltering: an open-label, cluster-randomized controlled trial. Am J Clin Nutr. 2017 Oct;106(4):1070-1077. doi: 10.3945/ajcn.117.157545. Epub 2017 Aug 23. PMID 28835364